CLINICAL TRIAL: NCT05669404
Title: Effects of the DASH and the Mediterranean Diet Combined With Salt Restriction on Blood Pressure Levels and Cardiometabolic Risk Factors in Adults With High Normal Blood Pressure or Grade 1 Hypertension: A Randomized Controlled Trial
Brief Title: Effects of the DASH vs. the Mediterranean Diet Combined With Salt Restriction on Blood Pressure Levels in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, MD, Ph.D., FESC, FACC, Professor of Cardiology, National and Kapodistrian University of Athens, Greece, Head of the First Cardiology Clinic, Hippocration General Hospital, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: The DASH-MedDiet study
Record Dates: First submitted 2022-12-14; First posted 2022-12-30 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Diet; Salt; Dietary Approaches to Stop Hypertension; Mediterranean; Dietary pattern
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Enrolled patients were blindly randomized with a 1:1:1:1 allocation to one of the four study groups, i.e., control group (CG), salt restriction group (SRG), DASH diet combined with salt restriction group (DDG), or MedDiet combined with salt restriction group (MDG).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of this study, which was a dietary intervention evaluating the effect of certain dietary strategies on blood pressure levels and cardiometabolic risk factors, masking of the trial participants and the clinical dietician (sub-investigator), who provided the dietary education and was solely responsible for the assignment of patients to the study groups was not possible. However, patients were completely unaware of the other groups of the study and were treated according to strict criteria, preventing deviations from the intended intervention. Moreover, the principal investigator, care providers, and all members of the medical team, who conducted the office and the ambulatory BP measurements (outcomes assessors) were blinded to patients' allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (CG) (No Intervention): Patients continued to consume their usual diet for 3 months
- Salt Restriction Group (SRG) (Experimental): Patients continued to consume their usual diet, but they restricted sodium intake to 2,000 mg/ day for 3 months.
  Interventions: Behavioral: Salt Restriction Group (SRG)
- DASH Diet combined with salt restriction Group (DDG) (Experimental): Patients consumed the DASH diet for 3 months.
  Interventions: Behavioral: DASH Diet combined with salt restriction Group (DDG)
- Mediterranean Diet combined with salt restriction Group (MDG) (Experimental): Patients consumed the MedDiet diet for 3 months.
  Interventions: Behavioral: Mediterranean Diet combined with salt restriction Group (MDG)

INTERVENTIONS:
Behavioral: Salt Restriction Group (SRG) — Patients assigned to the SRG continued to consume their usual diet, but they had to restrict their sodium intake to 2,000 mg/ day. They were given a detailed booklet containing information about table salt, foods rich in sodium, and practical ways to decrease salt consumption. During each 45-min individual session, they received intensive counselling and training to increase adherence to salt restriction. Also, they were instructed to keep their body weight stable and not to change their physical activity level over the next 3 months.
  Arms: Salt Restriction Group (SRG)
Behavioral: DASH Diet combined with salt restriction Group (DDG) — Patients assigned to the DDG received a more extensive booklet, which which in addition to the information regarding salt restriction, contained detailed information about the DASH diet, and practical advice about how to start and stay on the assigned dietary pattern. In addition to the booklet, each patient received an individualized eating plan with six sample daily menus, incorporating the goals of the DASH diet. During the 45-min individual sessions, patients were intensively counselled and trained to increase adherence to salt restriction and the assigned dietary pattern. Also, they were instructed to keep their body weight stable and not to change their physical activity level over the next 3 months.
  Arms: DASH Diet combined with salt restriction Group (DDG)
Behavioral: Mediterranean Diet combined with salt restriction Group (MDG) — Patients assigned to the MDG received a more extensive booklet, which which in addition to the information regarding salt restriction, contained detailed information about the MedDiet, and practical advice about how to start and stay on the assigned dietary pattern. In addition to the booklet, each patient received an individualized eating plan with six sample daily menus, incorporating the goals of the MedDiet diet. During the 45-min individual sessions, patients were intensively counselled and trained to increase adherence to salt restriction and the assigned dietary pattern. Also, they were instructed to keep their body weight stable and not to change their physical activity level over the next 3 months.
  Arms: Mediterranean Diet combined with salt restriction Group (MDG)

SUMMARY:
Non-pharmacological measures should serve as the first-line treatment in individuals with high normal blood pressure (BP) levels or grade 1 hypertension and low-moderate cardiovascular disease risk. Salt intake reduction and the dietary patterns of the Dietary Approaches to Stop Hypertension (DASH) diet and the Mediterranean diet (MedDiet) have been recognized as effective dietary measures for BP reduction. To the best of our knowledge, no clinical trials were designed to compare the effects of these dietary strategies. The purpose of the present trial was to compare the effects of salt restriction, the DASH, and the MedDiet combined with the salt restriction on BP levels and cardiometabolic risk factors in adults with high normal BP or grade 1 hypertension over 3 months.

DETAILED DESCRIPTION:
This was a 3-month, single-center, single-blind, randomized, controlled, clinical trial, with 4 parallel groups. Before their randomization, the potential participants visiting the Hypertension Unit of the Hippocration General Hospital of Athens for the first time were assessed for eligibility during two screen visits. Anthropometric measurements, demographic characteristics, dietary intake, physical activity level, smoking history, and alcohol consumption were recorded. In addition, office and ambulatory BP measurements, as well as fasting blood samples and 24-hour urine samples were obtained. Patients were eligible for inclusion if they had high normal BP (office systolic BP: 130-139 mmHg and/or office diastolic BP: 85-89 mmHg) or grade 1 hypertension (office systolic BP: 140-159 mmHg and/or office diastolic BP: 90-99 mmHg), based on the average of the means of the last two out of three measurements made during the two screen visits and were free of antihypertensive drug treatment and major medical conditions. Enrolled patients were blindly randomized to one of the four study groups, i.e., control group (CG), salt restriction group (SRG), DASH diet combined with salt restriction group (DDG), or MedDiet combined with salt restriction group (MDG). After randomization, all patients were followed monthly for 3 months in individual sessions, coordinated by the clinical dietician. For the patients of all four study groups, the goal was to maintain the initial body weight stable. Patients in the CG received the usual advice about salt restriction given to the patients by the clinical dietician at the Hypertension Unit. They were followed at the same frequency as the patients in the other study groups to obtain the study's intended measurements, without any other intervention. For the patients in the three intervention groups, the goal was to limit sodium intake to 2,000 mg/ day. Patients in the SRG were given a detailed booklet containing information about table salt and during each 45-min individual session, they received intensive counselling and training to increase adherence to salt restriction. Patients in the DDG and the MDG received a more extensive booklet, which also contained information about the assigned dietary pattern and an individualized eating plan, while during the 45-min individual sessions, patients in these two intervention groups were intensively counselled and trained to increase adherence to salt restriction and the assigned dietary pattern. Adherence to the assigned diet and/or salt restriction was established through subjective and objective measures, i.e., 7-day food records, adherence scores, and 24-hour urine tests. Anthropometric indices, dietary intake, physical activity level, and office BP were measured at baseline, and during each follow-up visit. Ambulatory BP measurements and collection of fasting blood samples and 24-hour urine samples were conducted at baseline and the end of the 3-month intervention.

ELIGIBILITY:
Inclusion Criteria:

1. High normal BP (office systolic BP: 130-139 mmHg and/or office diastolic BP: 85-89 mmHg) or grade 1 hypertension (office systolic BP: 140-159 mmHg and/or office diastolic BP: 90-99 mmHg) and low-moderate 10-year cardiovascular disease risk.
2. Willingness to participate in a dietary intervention to control BP and to attend individual sessions.
3. Signed informed consent form for participation.

Exclusion Criteria:

1. Current use of anti-hypertensive medications.
2. Current use of any other medications or agents affecting BP levels (e.g., nonsteroidal anti-inflammatory drugs).
3. Use of food supplements accompanied by a refusal to discontinue them.
4. Participation in a clinical study involving a drug or device within 3 months of screening.
5. Active weight loss or participation in a weight loss treatment program within 3 months of screening.
6. Secondary hypertension.
7. Atomic history of cardiovascular disease (e.g. acute myocardial infarction, stroke, heart failure).
8. Diabetes Mellitus (Type 1 & 2).
9. Chronic kidney disease, defined as an estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73m2.
10. Liver disease (e.g., hepatitis, cirrhosis).
11. Lung disease (e.g., chronic obstructive pulmonary disease).
12. Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
13. Celiac disease.
14. Active malignancy or cancer therapy.
15. Current major psychiatric disorder or current drug abuse.
16. Body Mass Index >40 kg/m2.
17. Current alcohol consumption >14 drinks per week.
18. Current or planned pregnancy before the end of the study, or breast-feeding.
19. Any concomitant conditions that in the opinion of the investigator interfere with the diet or other situations requiring specific nutritional management.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Office systolic blood pressure (BP) | 3 months post-intervention
  The attained mean office systolic BP difference among the randomized arms

SECONDARY OUTCOMES:
Office diastolic blood pressure (BP) | 3 months post-intervention
  The attained mean office diastolic BP difference among the randomized arms
Ambulatory systolic and diastolic blood pressure (BP) | 3 months post-intervention
  The attained between-group differences regarding the mean ambulatory BP measurements (during 24h, daytime, and night-time)
Odds of hypertension | 3 months post-intervention
  The odds of hypertension according to the office BP measurements in each study group
Metabolic syndrome and its components | 3 months post-intervention
  The attained between-group differences in metabolic syndrome presence and in the presence of individual metabolic syndrome components

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos P Tsioufis, Prof., Principal Investigator — First Cardiology Clinic, Hippocration General Hospital, NKUA
Locations (1):
- Hypertension Unit, First Cardiology Clinic, Hippocration General Hospital, National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No